CLINICAL TRIAL: NCT04281394
Title: Effects of Robot-assisted Gait Training in Patients Burn Injury on Lower Extremity : a Randomized Controlled Trial
Brief Title: Effects of Robot-assisted Gait Training in Patients Burn Injury on Lower Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-8
Record Dates: First submitted 2019-10-22; First posted 2020-02-24 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-10

CONDITIONS: Burns; Gait Disorder, Sensorimotor
Keywords: burns; rehabilitation; robot assisted gait training
MeSH Terms: conditions — Burns; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: patients with full or virtually full thickness involvement of >50% on the body surface area of the lower extremity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot assisted gait training (Experimental): Robot assisted gait training(RAGT) group received RAGT 5 sessions per week at duration 30 minutes with 30 minutes conventional physical therapy in 12 weeks. SUBAR® (CRETEM, Korea) is a wearable robot with a footplate that assists patients to perform voluntary muscle movements.
  Interventions: Device: Robot assisted gait training
- conventional physical training group (Active Comparator): The conventional group underwent conventional physical therapy( even level gait training and range of motion exercises) twice a day, 5 times a week in 12 weeks.
  Interventions: Other: conventional gait training

INTERVENTIONS:
Device: Robot assisted gait training — SUBAR® (CRETEM, Korea) is a wearable robot with a footplate that assists patients to perform voluntary muscle movements. RAGT group received RAGT 5 sessions per week at duration 30 minutes with 30 minutes conventional physical therapy in 12 weeks.
  Arms: Robot assisted gait training
Other: conventional gait training — even level gait training and range of motion exercises
  Arms: conventional physical training group

SUMMARY:
Gait enables individuals to move forward and is considered a natural skill. However, gait disturbances are very common in patients with burn injury. Major causes of functional impairment are pain and joint contractures. Recent studies focused on the application of robot-assisted gait training (RAGT). This study aimed to elucidate the efficacy and investigate the mechanism of motor recovery after RAGT on patients with lower extremity burn.

DETAILED DESCRIPTION:
This study aimed to elucidate the efficacy and investigate the mechanism of motor recovery after RAGT on patients with lower extremity burn.

20 patients with burn were randomly divided into 2 groups. RAGT group received RAGT 5 sessions per week at duration 30 minutes with 30 minutes conventional physical therapy in 12 weeks. SUBAR® (CRETEM, Korea) is a wearable robot with a footplate that assists patients to perform voluntary muscle movements. The conventional group underwent conventional physical therapy twice a day, 5 times a week in 12 weeks. Main outcomes were functional ambulatory category(FAC), 6 minutes walking test(6MWT), visual analogue scale(VAS), isometric forces of bilateral knee and ankle muscles, and foot pressure analysis before and after 12 weeks training.

ELIGIBILITY:
Inclusion Criteria:

* patients with full or virtually full thickness involvement of >50% on the body surface area of the lower extremity
* age > 18 years
* with ≤1 functional ambulation category (FAC) score ≤ 3

Exclusion Criteria:

* patients with cognitive disorders before burn
* serious cardiac dysfunction
* problems with weight bearing due to unstable fractures
* body weight ≥100 kg
* severe fixed contracture
* skin disorders that could be worsened by RAGT and conventional rehabilitation
* patients with severe pain who were unable to undergo conventional rehabilitation programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
the changes of functional ambulatory category | baseline, and after 12 weeks intervention
  Scale 0 means that the patient cannot walk or can only walk with assistance of two people. Scale 5 means that the patient can walk independently. Higher scores mean a better outcome.
the changes of 6 minutes walking test | baseline, and after 12 weeks intervention
  6MWT was performed in accordance with standardized guidelines, and the walking course was 20 m. Patients were instructed to walk as far as possible in 6 min. Higher scores mean a better outcome.
the changes of visual analogue scale | baseline, and after 12 weeks intervention
  Visual analogue scale was used to rate the degree of subjective pain during gait movement: 0 points were assigned when no pain was noted, and unbearable pain was assigned 10 points. higher scores mean a worse outcome

SECONDARY OUTCOMES:
the changes of active range of motion of flexion and extension | baseline, and after 12 weeks intervention
  The active range of motion(ROM) of different joints was measured using a goniometer and an inclinometer with a standardized technique(hip joint)
the changes of active range of motion of flexion and extension | baseline, and after 12 weeks intervention
  The active range of motion(ROM) of different joints was measured using a goniometer and an inclinometer with a standardized technique(knee joint)
the changes of active range of motion of dorsiflexion and plantarflexion | baseline, and after 12 weeks intervention
  The active range of motion(ROM) of different joints was measured using a goniometer and an inclinometer with a standardized technique(ankle joint)
the changes of isometric forces of knee flexion and knee extension | baseline, and after 12 weeks intervention
  Isometric knee extension and knee flexion muscle strength were measured by handheld dynamometer. Two measurements were taken using handheld dynamometer. Each trial lasted for 3-5 s, with 30 second rest period between trials. The higher of the two valid measurements was recorded.
the changes of isometric forces of ankle dorsiflexion and ankle plantarflexion | baseline, and after 12 weeks intervention
  Isometric ankle dorsiflexion, and ankle plantar flexion muscle strength were measured by handheld dynamometer. Two measurements were taken using handheld dynamometer. Each trial lasted for 3-5 s, with 30 second rest period between trials. The higher of the two valid measurements was recorded.
the changes of gait symmetry using stride length | baseline, and after 12 weeks intervention
  Stride is the equivalent of a gait cycle. The duration of a stride is the interval between two sequential initial floor contacts by the same limb. symmetry ratio is defined with affected side stride length/ non affected side stride length.
the changes of center of foot pressure pattern | baseline, and after 12 weeks intervention
  center of foot pressure patten during a normal stride. longitudinal line analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goto K, Morishita T, Kamada S, Saita K, Fukuda H, Shiota E, Sankai Y, Inoue T. Feasibility of rehabilitation using the single-joint hybrid assistive limb to facilitate early recovery following total knee arthroplasty: A pilot study. Assist Technol. 2017 Winter;29(4):197-201. doi: 10.1080/10400435.2016.1219883. Epub 2016 Aug 10. PMID 27689789
- [Result] Kang MG, Yun SJ, Shin HI, Kim E, Lee HH, Oh BM, Seo HG. Effects of robot-assisted gait training in patients with Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2019 Jan 7;20(1):15. doi: 10.1186/s13063-018-3123-4. PMID 30616685